CLINICAL TRIAL: NCT06426823
Title: The Role of GIP in Postprandial Splanchnic Blood Flow Distribution and Metabolism in Patients With Type 2 Diabetes
Acronym: GA-17b
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: GA-17b
Record Dates: First submitted 2024-05-06; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Blood Flow
Keywords: Gut hormones; GIP; Physiology; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Single blind, placebo controlled, randomized, crossover study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Saline and oral water (SAL-WAT) (Placebo Comparator): Saline infusion, oral water ingestion
  Interventions: Other: Saline / placebo
- Saline infusion and oral glucose ingestion (SAL-GLU) (Active Comparator): Saline infusion, oral glucose ingestion
  Interventions: Other: Saline / placebo
- GIP(3-30)NH2 infusion and oral water ingestion (GIA-WAT) (Experimental): GIPR antagonist infusion, oral water ingestion
  Interventions: Other: GIPR antagonist / study tool
- GIP(3-30)NH2 infusion and oral glucose ingestion (GIA-GLU) (Experimental): GIPR antagonist infusion, oral glucose ingestion
  Interventions: Other: GIPR antagonist / study tool

INTERVENTIONS:
Other: Saline / placebo — NaCl (9 mg/ml)
  Arms: Saline and oral water (SAL-WAT); Saline infusion and oral glucose ingestion (SAL-GLU)
Other: GIPR antagonist / study tool — GIP(3-30)NH2
  Arms: GIP(3-30)NH2 infusion and oral glucose ingestion (GIA-GLU); GIP(3-30)NH2 infusion and oral water ingestion (GIA-WAT)

SUMMARY:
This project will describe the mechanisms of action and the relative contributions of GIP to changes in gastrointestinal blood flow induced by oral glucose and endogenous GIP with the use of a receptor antagonists GIP(3-30)NH2 in patients with type 2 diabetes.

DETAILED DESCRIPTION:
Each participant will attend four independent randomised experimental days in the MRI-scanner with intravenous infusion (hormone/placebo) and oral ingestion (glucose/water): An intravenous infusion of saline or GIP(3-30)NH2 starts at time point -20 minutes.The infusions are combined with an oral glucose tolerance test (75 gram of glucose dissolved in 250 ml water ingested orally) at time point 0 minutes on two of the experimental days (with and without GIP(3-30)NH2).

MRI measurements are repeatedly performed and blood samples are drawn to be analysed for endocrine responses from the intestines, pancreas, and bones.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* BMI 20-35 kg/m^2
* Age 20-80

Exclusion Criteria:

* Not MRI-compatible implants
* Claustrophobia
* Abnormal kidney or liver function
* Anemia
* Planned weight loss or change in diet
* Hypertension
* Other conditions that could be expected to affect the primary or secondary outcomes

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Redistribution of splanchnic blood flow in the vessel mesenteric superior artery (functional MRI) | 80 minutes
  Measued with phase-contrast MRI in ml/min

SECONDARY OUTCOMES:
GIP levels | 80 minutes
  Radioimmuno assay on plasma blood sample (pmol/L)
GIP(3-30)NH2 levels | 80 minutes
  Radioimmuno assay on plasma blood sample (nmol/L)
Glucose | 80 minutes
  Bedside measurement of whole blood sample (mmol/L)
C-peptide | 80 minutes
  Electrochemiluminescence immunoassay of plasma blood sample (pmol/L)
Insulin | 80 minutes
  Electrochemiluminescence immunoassay of plasma blood sample (pmol/L)
Glucagon | 80 minutes
  Radioimmuno assay on plasma blood samples (pmol/L)
Blood flow in portal vein | 80 minutes
  Measued with phase-contrast MRI in ml/min
Blood flow in coeliac trunc | 80 minutes
  Measued with phase-contrast MRI in ml/min
Blood flow in hepatic artery | 80 minutes
  Measued with phase-contrast MRI in ml/min

CONTACTS AND LOCATIONS:
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Will share upon requests

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-17): https://cdn.clinicaltrials.gov/large-docs/23/NCT06426823/Prot_SAP_000.pdf